CLINICAL TRIAL: NCT05711537
Title: Auricular Acupressure as a Non-Opioid Adjuvant in Opioid Tolerant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00068022
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use Disorder
Keywords: Chronic Pain; Opioid Use Disorder; Acupressure
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Any patient admitted to Atrium Health Wake Forest Baptist for which our chronic pain/addiction medicine service is consulted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Auricular Acupressure (AA) Group (Experimental): Participants will participate in the Auricular Acupressure intervention over 3 days in addition to the Standard of Care treatment for Chronic Pain and complete questionnaires
  Interventions: Device: Auricular Acupressure with Vaccaria 600t ear seeds

INTERVENTIONS:
Device: Auricular Acupressure with Vaccaria 600t ear seeds — Auricular Acupressure utilizing vaccaria 600 t ear seeds applied to 5 designated sites to each ear. Both ears will have seeds applied. Participants will be asked if they consent to having their intervention session photographed and audio recorded in collaboration with the BAA press training and intervention fidelity study.
  Other Names: vaccaria 600 t ear seeds

SUMMARY:
The purpose of this study is to determine if the addition of auricular acupressure to the typical pharmacological regimen given to patients on the chronic pain/addiction service will lower pain scores and decrease pain medication usage.

DETAILED DESCRIPTION:
Participants will be asked to complete baseline questionnaires. After completion, a study interventionist will place 10 adhesive acupressure pads./seeds on the participant's ears, 5 acupressure pads per ear. The pads will be placed on specific sites of the ear that are thought to help with pain and overall well-being. Over the course of 3 days, participants will be asked to apply a small amount of pressure with their finger to each of the pads and answer study questionnaires.

This feasibility trial is being performed in collaboration with the Battlefield Auricular Acupressure (BAApress) Training and Intervention Fidelity study (IRB00084011).

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18
* History of documented chronic pain with or without opioid use disorder (Polysubstance abuse or opioid use disorder or opioid narcotic use documented as home medication)
* Estimated length of stay (admission) at least 5 days at the time of recruitment
* Able to read and understand informed consent form

Exclusion Criteria:

* Patient refusal
* Patients with a known history of leaving against medical advice (AMA)
* only English-speaking participants will be eligible.
* Inability to communicate via telephone
* Participants with a history of skin disease (e.g., psoriasis) involving the ear, adhesive allergy, recent scar tissue on ear, or current abrasions or cuts on ear,
* Cognitive impairment (delirium, dementia)
* Physical impairment preventing them from applying pressure to the beads
* Patients with cardiac pacemakers (contraindication to POINTER PAL)
* Use of some types of hearing aids (obstructing the placement of beads)
* Any chronic or acute illness or psychiatric conditions that would impact adherence to the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Columbano, M.D., Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Auricular Acupressure (AA) Group
Started | 21
Completed | 18
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Using Numerical Rating Scale (NRS)
Description: In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale | 6.62 (1.36)

2. Primary Outcome: Pain Scores Using Numerical Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Day 1
Population: 1 subject withdrew participation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 20
score on a scale | 7 (1.86)

3. Primary Outcome: Pain Scores Using Numerical Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Day 2
Population: 1 subject withdrew after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 20
score on a scale | 7.2 (2.22)

4. Primary Outcome: Pain Scores Using Numerical Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Day 3
Population: 1 subject withdrew after baseline and 2 were discharged home on day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 18
score on a scale | 6.68 (2.26)

5. Primary Outcome: Pain, Enjoyment and General Activity (PEG) Assessment Scores
Description: Patient reported assessment of pain intensity and interference. We will compare scores before and after initiation of Auricular Acupressure.
  The PEG scale consists of 3 separate numerical scales: PEG-1 What number best describes your pain this week?, PEG-2 What number describes how during the past week pain has interfered with your enjoyment of life?, and PEG-3 What number best describes how during the past week pain has interfered with your general activity?
  Each scale has ratings ranging from 0-10. Individuals rate their pain level concerning 3 different areas. Higher scores represent more pain and or increased enjoyment and activity interference.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale
  PEG-1 | 7 (1.76)
  PEG-2 | 7.57 (2.36)
  PEG-3 | 7.71 (2.45)

6. Primary Outcome: Pain, Enjoyment and General Activity (PEG) Assessment Scores
Description: as for outcome 5
Time Frame: Day 3
Population: 1 withdrew study participation after day 1 and 2 were discharged home
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 18
score on a scale
  PEG-1 | 6.5 (1.86)
  PEG-2 | 5.89 (3.03)
  PEG-3 | 6.44 (3.22)

7. Primary Outcome: Visual Analogue Scale (VAS)
Description: Scores range from 0-100. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale | 65.85 (17.71)

8. Secondary Outcome: Changes in Amount of Opioid Use
Description: Pre-Admission Opioid requirement and change from baseline (medication used during the intervention and as reported afterwards vs. home dose before the study started) collecting type, frequency and milligram use and date and time of last use prior to admission measuring mean/median changes from Baseline to Day 3 post evaluation.
Time Frame: Baseline, Day 1, Day 2, and Day 3
Population: morphine mg equivalents (MME) total excluding buprenorphine
Measure: Mean (Standard Error); unit: morphine mg equivalents
Groups:
- Intervention Auricular Acupressure (AA) Group-Baseline; Intervention Auricular Acupressure (AA) Group-DAY 1; Intervention Auricular Acupressure (AA) Group-DAY 2; Intervention Auricular Acupressure (AA) Group-DAY 3: Participants will participate in the Auricular Acupressure intervention over 3 days in addition to the Standard of Care treatment for Chronic Pain and complete questionnaires
  Auricular Acupressure with Vaccaria 600t ear seeds: Auricular Acupressure utilizing vaccaria 600 t ear seeds applied to 5 designated sites to each ear. Both ears will have seeds applied. Participants will be asked if they consent to having their intervention session photographed and audio recorded in collaboration with the BAA press training and intervention fidelity study.
Arm/Group | Intervention Auricular Acupressure (AA) Group-Baseline | Intervention Auricular Acupressure (AA) Group-DAY 1 | Intervention Auricular Acupressure (AA) Group-DAY 2 | Intervention Auricular Acupressure (AA) Group-DAY 3
Number analyzed (Participants) | 21 | 20 | 20 | 18
morphine mg equivalents | 84.95 (46.14) | 67.34 (19.88) | 71.01 (22.62) | 53.16 (19.14)

9. Secondary Outcome: Willingness to Decrease Dependence Scores
Description: Assessment of patient's willingness or desire to decrease opioid dependence and usage will be assessed by asking the subject to answer (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree - A higher score denotes a greater willingness to decrease dependence.
Time Frame: Day 3
Population: percentage of total subjects who desire to decrease their dependency on opioids: answer as strongly disagree, neither agree or disagree, agree, or strongly agree
Measure: Number; unit: percentage of participants
Groups:
- Strongly Disagree: I want to decrease my dependency on opioids:
  Strongly disagree
- Neither Agree or Disagree: I want to decrease my dependency on opioids:
  Neither agree or disagree
- Agree: I want to decrease my dependency on opioids:
  Agree
- Strongly Agree: I want to decrease my dependency on opioids:
  Strongly agree
Arm/Group | Strongly Disagree | Neither Agree or Disagree | Agree | Strongly Agree
Number analyzed (Participants) | 18 | 18 | 18 | 18
percentage of participants | 15.79 | 26.32 | 21.05 | 36.84

10. Secondary Outcome: Generalized Anxiety Disorder (GAD-7) Score Changes
Description: A 7 item scale to identify Generalized Anxiety Disorder symptoms of evaluation. Patients are asked to rate anxiety symptoms on a scale of 0-3. Total scores for all 7 items range from 0-21. Higher scores indicate increased severity.
Time Frame: Baseline and Day 3
Population: 17 paired assessments on Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline; DAY 3: Participants will participate in the Auricular Acupressure intervention over 3 days in addition to the Standard of Care treatment for Chronic Pain and complete questionnaires
  Auricular Acupressure with Vaccaria 600t ear seeds: Auricular Acupressure utilizing vaccaria 600 t ear seeds applied to 5 designated sites to each ear. Both ears will have seeds applied. Participants will be asked if they consent to having their intervention session photographed and audio recorded in collaboration with the BAA press training and intervention fidelity study.
Arm/Group | Baseline | DAY 3
Number analyzed (Participants) | 21 | 17
score on a scale | 10.9 (5.3) | 9.53 (6.12)

11. Secondary Outcome: Pain Catastrophizing Scale (PCS) Assessments
Description: The assessment of thoughts and feelings of the patients will be assessed using questions that are rated 0 for not at all to 4 for all the time. "The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking due to low back pain according to 3 components: rumination, magnification, and helplessness. It is a 13-item scale, with a total range of 0 to 52. Higher scores are associated with higher amounts of pain catastrophizing."
Time Frame: Baseline and Day 3
Population: 16 paired assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | DAY 3
Number analyzed (Participants) | 21 | 17
score on a scale | 23.15 (13.83) | 24.82 (13.39)

12. Secondary Outcome: Auricular Acupressure Acceptability-DAY 3-Satisfaction
Description: Three questions were asked to evaluate acceptance of the intervention (Auricular Acupressure) the first was a Likert scale satisfaction question. This outcome pertains only to the following acceptability question: "How satisfied were you with how your pain has been treated?" using the Likert scale to measure "Very satisfied =5, Satisfied=4, Somewhat satisfied = 3, Somewhat dissatisfied= 2, Dissatisfied 1, Very Dissatisfied 0
Time Frame: Day 3
Measure: Number; unit: percentage of participants
Groups:
- DAY 3-Satisfaction: acceptability questions: "How satisfied were you with how your pain has been treated?" using the Likert scale to measure "Very satisfied =5, Satisfied=4, Somewhat satisfied = 3, Somewhat dissatisfied= 2, Dissatisfied 1, Very Dissatisfied 0
Arm/Group | DAY 3-Satisfaction
Number analyzed (Participants) | 19
percentage of participants
  Answered "Very Satisfied" | 21.05
  Answered "Satisfied" | 21.05
  Answered "Somewhat satisfied" | 47.4
  Answered "Dissatisfied" | 10.5

13. Secondary Outcome: Auricular Acupressure Acceptability--DAY 3-future Use
Description: Three questions were asked to evaluate acceptance of the intervention (Auricular Acupressure). The second question posed a yes/no question. This outcome pertains only to the following question:
  Would you consider using auricular acupressure in the future for pain or if recommended by your nurse or physician? a. No, would not use again (Score of 0) b. Maybe (Score of 1), c. Yes, I would consider using in the future (Score of 2) 3
Time Frame: Day 3
Measure: Number; unit: Percentage of participants
Groups:
- DAY 3-future Use: Would you consider using auricular acupressure in the future for pain or if recommended by your nurse or physician? a. No, would not use again (Score of 0) b. Maybe (Score of 1), c. Yes, I would consider using in the future (Score of 2) 3
Arm/Group | DAY 3-future Use
Number analyzed (Participants) | 19
Percentage of participants
  Answered "No, would not use again" | 15.8
  Answered "Maybe" | 31.6
  Answered "Yes, would definitely consider using again" | 52.6

14. Secondary Outcome: Change in Patient Global Impression of Change (PGIC) Scores
Description: Patient reported assessment of improvement or decline of their pain - The patient enters his answer on a 7-point scale scored as: (1) "very much better," (2) "much better," (3) "a little better," (4) "no change," (5) "a little worse," (6) "much worse," or (7) "very much worse."
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline-PGIC; DAY 3-PGIC: Patient reported assessment of improvement or decline in their pain.
Arm/Group | Baseline-PGIC | DAY 3-PGIC
Number analyzed (Participants) | 18 | 18
score on a scale | 3.33 (.686) | 3.22 (.878)

15. Secondary Outcome: Changes in Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: Sleep disturbance is a patient reported assessment on the quality of their sleep - Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline-PROMIS; DAY 3-PROMIS: Patient reported assessment of sleep disturbance.
Arm/Group | Baseline-PROMIS | DAY 3-PROMIS
Number analyzed (Participants) | 21 | 18
score on a scale | 21.85 (5.62) | 17.89 (6.32)

16. Other Pre Specified Outcome: Auricular Acupressure Acceptability--Qualitative Question
Description: Three questions were asked to evaluate acceptance of the intervention (Auricular Acupressure). The third question was a qualitative question: "Is there anything else you would like to tell us that may be helpful for us to know regarding ear acupressure?
Time Frame: Day 3
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Battlefield Auricular Acupressure (BAApress)
Description: The Interventionist's (Acupressure nurse) will be asked to capture time related to completion of study tasks and other qualitative questions to assess overall feasibility.
Time Frame: Day 1
Reporting Status: Not Posted

18. Primary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 7
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale | 65.42 (28.08)

19. Primary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 7
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale | 70.10 (25.91)

20. Primary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 7
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Auricular Acupressure (AA) Group
Number analyzed (Participants) | 21
score on a scale | 70.05 (29.31)

ADVERSE EVENTS:
Time Frame: adverse events reported over 3 days
Arm/Group | Intervention Auricular Acupressure (AA) Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT05711537/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT05711537/ICF_000.pdf